CLINICAL TRIAL: NCT05433454
Title: Outreach and Maintenance of Medicaid Enrollment: Evidence From Wisconsin's Navigator Program
Brief Title: Impact of Outreach on Medicaid Enrollment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Covering Wisconsin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0806; Protocol Amend 2/21/2024 (Other: UW Madison); A538500 (Other: UW Madison); SMPH/POP HEALTH SCI/POP HLTH (Other: UW Madison)
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Health Insurance
Keywords: Outreach; Enrollment; Medicaid

STUDY DESIGN:
Intervention Model Description: The nature of the intervention will be randomized to participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Outreach via Postcard (Experimental): 40 percent of the sample
  Interventions: Other: Outreach From Navigators
- Outreach via Postcard + Outbound Call (Experimental): Outreach via postcard, plus placed an outbound phone call from navigators (20% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach via Text Message Encouraging Call to Hotline (Experimental): Outreach via text message encouraging a call to a hotline for assistance (15% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach via Text Message Encouraging Call to Hotline + Outbound Call (Experimental): Outreach via text message encouraging a call to a hotline for assistance, plus outbound phone call from navigators (7.5% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach via Text Message Encouraging Text Reply To Connect with Navigators (Experimental): Outreach via text message encouraging a text reply to connect with navigators via chatbot (15% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach via Text Message Encouraging Text Reply To Connect with Navigators + Outbound Call (Experimental): Outreach via text message encouraging a text reply to connect with navigators via chatbot, plus an outbound phone call from navigators (7.5% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach via Text Message Encouraging a Call to a Hotline for Assistance + a Reminder Message (Experimental): Outreach via text message encouraging a call to a hotline for assistance plus a similar reminder message two weeks later (15% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach Text Message Encouraging Call a Hotline for Assistance + Reminder Message (Experimental): Outreach via text message encouraging a call to a hotline for assistance plus a similar reminder message two weeks later + outbound call (7.5% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach via Text Message Encouraging Text Reply To Connect with Navigators+ a Reminder Message (Experimental): Outreach via text message encouraging a text reply to connect with navigators via chatbot plus a similar reminder message two weeks later (15% of sample)
  Interventions: Other: Outreach From Navigators
- Outreach via Text Message Encouraging Reply To Connect with Navigators + Reminder Message (Experimental): Outreach via text message encouraging a text reply to connect with navigators via chatbot plus a similar reminder message two weeks later + outbound call (7.5% of sample)
  Interventions: Other: Outreach From Navigators

INTERVENTIONS:
Other: Outreach From Navigators — Navigators are professionals who can provide one-on-one assistance with the Medicaid renewal process. The nature of the outreach will be randomized to participants.

SUMMARY:
This project will assess the impact of various forms of outreach from navigators on Medicaid enrollment. Navigators are professionals who can provide one-on-one assistance with the Medicaid renewal process. The investigators propose to randomize the nature of outreach to households in Wisconsin enrolled in fee-for-service Medicaid who must renew or lose their coverage.

DETAILED DESCRIPTION:
During the COVID-19 public health emergency, states received support to maintain continuous Medicaid coverage, raising Medicaid enrollment to unprecedented levels. In Wisconsin, enrollment was nearly 30% higher by the end of 2021 compared to February 2020, with the maintenance of enrollment policy contributing to much of this increase. After the end of the public health emergency, normal renewal processes will resume.

The Wisconsin navigator program, Covering Wisconsin, has been commissioned by the Department of Health Services (DHS) to conduct outreach to the group of fee-for-service Medicaid beneficiaries who need to re-determine eligibility after the conclusion of the public health emergency. To identify what outreach strategies are most effective, the investigators propose to randomize the nature of outreach used. While there will be some variation in the content and timing of messages, all beneficiaries will receive messages with clear information on how to contact the navigators.

Per a protocol amendment approved on 2/21/24, the study team will no longer randomize receipt of an outbound call but rather will provide it to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Included on the lists Wisconsin DHS provides to Covering Wisconsin of fee-for-service Medicaid beneficiaries who need to renew their Medicaid coverage

Exclusion Criteria:

* Prefer a language other than English or Spanish or lack a cellular phone number

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 119308 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Renew Medicaid Coverage | up to 1 year

OTHER OUTCOMES:
Number of Participants Who Submit an Application to Renew Medicaid Coverage | up to 1 year
Number of Participants for Whom Application to Renew Medicaid Coverage is Denied for Administrative Reasons | up to 1 year
Demographics of People who Renew Medicaid Coverage | up to 1 year
  The investigators will measure the characteristics of people who renew medicaid coverage, including baseline income, race/ethnicity, and language preference.
Number of Participants Responding 'DONE' to Text Message Outreach | up to 1 year
Survey of Participants Who Received an Outbound Call Reported in Count of Participants | up to 1 year
  People who received an outbound call will be asked whether they finished an application to renew their coverage or receive new coverage, and whether they received a text message or postcard with a reminder and information about how to get help.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Myerson, MPH, PhD, Principal Investigator — UW-Madison School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No